CLINICAL TRIAL: NCT00775645
Title: S0715: Randomized Placebo-Controlled Trial of Acetyl-L-Carnitine (ALC) for the Prevention of Taxane Induced Neuropathy Phase III
Brief Title: S0715: Acetyl-L-Carnitine in Preventing Neuropathy in Women With Stage I, II, or IIIA Breast Cancer Undergoing Chemo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000617081; S0715 (Other: SWOG); U10CA037429 (NIH)
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer; Chemotherapeutic Agent Toxicity; Fatigue; Neuropathy; Neurotoxicity
Keywords: neurotoxicity; chemotherapeutic agent toxicity; fatigue; neuropathy; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Neurotoxicity Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive oral acetyl-L-carnitine hydrochloride 3 times daily for 24 weeks.
  Interventions: Dietary Supplement: acetyl-L-carnitine hydrochloride
- Arm II (Placebo Comparator): Patients receive oral placebo 3 times daily for 24 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: acetyl-L-carnitine hydrochloride — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Acetyl-L-carnitine may prevent or lessen neuropathy caused by chemotherapy. It is not yet known whether acetyl-L-carnitine is more effective than a placebo in preventing neuropathy caused by chemotherapy.

PURPOSE: This randomized phase III trial is studying acetyl-L-carnitine to see how well it works compared with a placebo in preventing neuropathy in women with stage I, stage II, or stage III breast cancer undergoing chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare whether treatment with acetyl-L-carnitine hydrochloride vs placebo prevents symptoms of neuropathy as measured by the 11-item neurotoxicity component of the FACT-Taxane Questionnaire at 12 weeks after study registration in women with stage I, II, or IIIA breast cancer undergoing adjuvant taxane-based chemotherapy.

Secondary

* Compare the functional status of these patients using the Trial Outcome Index from the Functional Assessment of Cancer Therapy (FACT)-Taxane Questionnaire.
* Compare fatigue in these patients using the Function Assessment of Chronic Illness Therapy (FACIT)-Fatigue Symptom Module.

Other

* Compare the proportion of patients experiencing grade 3 or 4 neuropathy.
* Compare serum nerve growth factor levels in these patients.
* Describe the total dose of taxane received and treatment delays, compliance with therapy, and use of concurrent medications, dietary supplements (e.g., glutamine), vitamin E, and complementary and alternative medicines in these patients.
* Explore the relationship between nerve growth factor levels and the degree of neuropathy and functional status in these patients.
* Explore the relationship between genetic markers responsible for taxane metabolism and clearance (e.g., CYP2C8, CYP3A4, CYP3A5, GSTM1, and GSTP1) and the degree of neuropathy in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to planned adjuvant chemotherapy regimen for breast cancer (paclitaxel weekly for 12 weeks vs paclitaxel biweekly for 4 courses [8 weeks] vs paclitaxel biweekly for 6 courses [12 weeks] vs docetaxel every 3 weeks for 4 courses [12 weeks] vs docetaxel every 3 weeks for 6 courses [18 weeks]) and age (< 60 years vs ≥ 60 years). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral acetyl-L-carnitine hydrochloride 3 times daily for 24 weeks.
* Arm II: Patients receive oral placebo 3 times daily for 24 weeks. Patients complete the FACT-Taxane Trial Outcome Index and the FACIT-Fatigue Symptom Module questionnaires at baseline, at 12, 24, and 36 weeks, and at 1 and 2 years.

Blood samples are collected at baseline and at week 12 for biomarker analysis (nerve growth factor levels) by ELISA, DNA extraction, and genotyping analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary invasive adenocarcinoma of the breast

  * Stage I-III disease
  * No metastatic disease
* Must have undergone modified radical mastectomy or breast-sparing surgery
* Planning to receive one of the following standard taxane-based systemic chemotherapy regimens as adjuvant therapy for breast cancer:

  * Paclitaxel 80 mg/m² weekly for 12 weeks
  * Paclitaxel 175 mg/m² every other week for 4 courses (8 weeks)
  * Paclitaxel 175 mg/m² every other week for 6 courses (12 weeks)
  * Docetaxel 75 mg/m² every 3 weeks for 4 courses (12 weeks)
  * Docetaxel 75 mg/m² every 3 weeks for 6 courses (18 weeks)
* No history of neuropathy
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Zubrod performance status 0-2
* Serum creatinine ≤ 2.5 times upper limit of normal
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Able to complete questionnaires in English or Spanish
* Willing to submit blood samples for DNA extraction, genotyping analysis, and nerve growth factor studies
* No history of diabetes
* No history of seizure disorder
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, ductal carcinoma in situ, or adequately treated stage I or stage II malignancy from which the patient is currently in complete remission

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior breast surgery
* Prior neoadjuvant or adjuvant chemotherapy allowed
* No prior taxane therapy
* No prior biologic therapy for treatment of breast cancer
* No concurrent vitamin E, glutamine, gabapentin, nortriptyline, amitriptyline, or duloxetine hydrochloride

  * Multivitamins containing vitamin E allowed provided vitamin E dose is < 1,000 IU
* No concurrent anti-seizure medications
* Concurrent hormonal therapy allowed
* Concurrent biologic therapy allowed (e.g., Herceptin)
* Concurrent participation in another therapeutic clinical trial allowed

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence H. Baker, DO, FACOI, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (295):
- United States (295):
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Providence Cancer Center, Anchorage, Alaska
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Valley Medical Oncology, Fremont, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Sutter Health - Western Division Cancer Research Group, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center - Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente - Denver, Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Kaiser Permanente - Lafayette, Lafayette, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Cancer Care at Our Lady of Bellefonte Hospital, Ashland, Kentucky
  - Northeast Louisiana Cancer Institute at St. Francis Medical Center, Alexandria, Louisiana
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Lapeer Regional Hospital, Lapeer, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Skaggs Cancer Center at Skaggs Regional Medical Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Presbyterian Cancer Treatment Center at Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center - South, Las Cruces, New Mexico
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Cleveland Clinic Beachwood Family Health and Surgery Center, Beachwood, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - St. Charles Medical Center - Bend, Bend, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Northwest Cancer Specialists at Rose Quarter Cancer Center, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - AnMed Cancer Center, Anderson, South Carolina
  - Cancer Centers of the Carolinas - Easley, Easley, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Self Regional Cancer Center at Self Regional Medical Center, Greenwood, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Pacific Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Legacy Salmon Creek Medical Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hershman DL, Unger JM, Crew KD, Minasian LM, Awad D, Moinpour CM, Hansen L, Lew DL, Greenlee H, Fehrenbacher L, Wade JL 3rd, Wong SF, Hortobagyi GN, Meyskens FL, Albain KS. Randomized double-blind placebo-controlled trial of acetyl-L-carnitine for the prevention of taxane-induced neuropathy in women undergoing adjuvant breast cancer therapy. J Clin Oncol. 2013 Jul 10;31(20):2627-33. doi: 10.1200/JCO.2012.44.8738. Epub 2013 Jun 3. PMID 23733756

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 437 accrued patients, 27 were ineligible and 1 withdrew consent.
Groups:
- Arm I (Acetyl-L-carnitine Hydrochloride)): Patients receive oral acetyl-L-carnitine hydrochloride 3 times daily for 24 weeks
- Arm II (Placebo): Patients receive oral placebo 3 times daily for 24 weeks
Period: Overall Study
Arm/Group | Arm I (Acetyl-L-carnitine Hydrochloride)) | Arm II (Placebo)
Started | 208 | 201
Completed | 191 | 181
Not Completed | 17 | 20

BASELINE CHARACTERISTICS:
Population: 437 patients registered, 27 ineligible, 1 withdrew consent, 409 evaluable patients at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Acetyl-L-carnitine Hydrochloride)) | Arm II (Placebo) | Total
Number analyzed (Participants) | 208 | 201 | 409
Age, Continuous [Median (Full Range); unit: years] | 52 [27 to 80] | 50 [26 to 77] | 52 [26 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 208 | 201 | 409
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 15 | 36
  Not Hispanic or Latino | 181 | 177 | 358
  Unknown or Not Reported | 6 | 9 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 12 | 8 | 20
  Native Hawaiian or Other Pacific Islander | 4 | 2 | 6
  Black or African American | 17 | 20 | 37
  White | 160 | 165 | 325
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 12 | 5 | 17
Zubrod Performance Status [Count of Participants; unit: Participants] — 0 - Asymptomatic (Fully active, able to carry on all predisease activities without restriction)
  1. - Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. - Symptomatic, <50% in bed during the day (Ambulatory and capable of all self care but unable to carry out any work activities.
  Participants
    0 | 156 | 146 | 302
    1 | 51 | 54 | 105
    2 | 1 | 1 | 2
Breast cancer stage [Count of Participants; unit: Participants] — As per AJCC 6th ed, 2002:
  https://cancerstaging.org/references-tools/deskreferences/Documents/AJCC6thEdCancerStagingManualPart2.pdf
  Participants
    I | 57 | 50 | 107
    II | 110 | 107 | 217
    III | 41 | 43 | 84
    Not measurable/measured | 0 | 1 | 1
Taxane regiment [Count of Participants; unit: Participants]
  Paclitaxel | 124 | 123 | 247
  Docetaxel | 84 | 77 | 161
  Not measurable/measured | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: 12-week FACT-Taxane Neurotoxicity Model-adjusted Score in ALC and Placebo Groups
Description: Compare whether treatment with acetyl-L-carnitine hydrochloride vs placebo prevents symptoms of neuropathy as measured by the 11-item neurotoxicity (NTX) component of the Functional Assesment of Cancer Therapy (FACT)-Taxane Questionnaire at 12 weeks after study registration in women with breast cancer undergoing adjuvant taxane-based chemotherapy. Linear regression model adjusted for baseline score, taxane regiment, and age. Lower scores indicate worse CIPN. Total possible range is 0 to 64. For more information on this subscale, please see http://www.facit.org/FACITOrg/Questionnaires
Time Frame: 12 weeks post-registration
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Arm I (Acetyl-L-carnitine Hydrochloride)) | Arm II (Placebo)
Number analyzed (Participants) | 191 | 181
units on a scale | 35.4 [34.1 to 36.7] | 36.3 [35 to 37.6]
Statistical Analysis 1: Comparison: Arm I (Acetyl-L-carnitine Hydrochloride)) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.17, Regression, Linear; Linear regression model adjusted for baseline score, taxane regiment, and age; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-2.2 to 0.4]

2. Secondary Outcome: 12-week FACT-Trial Outcome Index(TOI) Functional Status Model-adjusted Score in ALC and Placebo Groups
Description: Compare FACT-TOI outcome in treatment vs placebo groups at 12 weeks after study registration in women with breast cancer undergoing adjuvant taxane-based chemotherapy. Linear regression model adjusted for baseline score, taxane regiment, and age. Lower scores indicate worse functional status. Total possible range is 0 to 120. For more information on this subscale, please see http://www.facit.org/FACITOrg/Questionnaires
Time Frame: 12 weeks post-registration
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Arm I (Acetyl-L-carnitine Hydrochloride)) | Arm II (Placebo)
Number analyzed (Participants) | 191 | 181
units on a scale | 92.1 [89.3 to 94.9] | 92.3 [89.4 to 95.1]
Statistical Analysis 1: Comparison: Arm I (Acetyl-L-carnitine Hydrochloride)) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.92, Regression, Linear; Linear regression model adjusted for baseline score, taxane regiment, and age; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-3 to 2.7]

3. Secondary Outcome: 12-week FACIT-fatigue Model-adjusted Score in ALC and Placebo Groups
Description: Compare fatigue outcome between treatment and placebo groups as measured by the 13-item Functional Assessment of Chronic Illness Therapy FACIT-fatigue questionnaire at 12 weeks after study registration in women with breast cancer undergoing adjuvant taxane-based chemotherapy. Linear regression model adjusted for baseline score, taxane regiment, and age. Lower scores indicate more fatigue. Total possible range is 0 to 52. For more information on this subscale, please see http://www.facit.org/FACITOrg/Questionnaires
Time Frame: 12 weeks post-registration
Measure: Mean (Full Range); unit: FACIT-fatigue score
Arm/Group | Arm I (Acetyl-L-carnitine Hydrochloride)) | Arm II (Placebo)
Number analyzed (Participants) | 191 | 181
FACIT-fatigue score | 36.6 [34.7 to 38.6] | 35.3 [33.4 to 37.3]
Statistical Analysis 1: Comparison: Arm I (Acetyl-L-carnitine Hydrochloride)) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.20, Regression, Linear; Linear regression model adjusted for baseline score, taxane regiment, and age; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-0.7 to 3.3]

4. Other Pre Specified Outcome: Proportion of Patients Experiencing Grade 3 or 4 Neuropathy
Description: Proportion of patients experiencing grade 3 or 4 neuropathy
Time Frame: 12 weeks post-registration
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Acetyl-L-carnitine Hydrochloride)) | Arm II (Placebo)
Number analyzed (Participants) | 202 | 194
Participants | 8 | 1
Statistical Analysis 1: Comparison: Arm I (Acetyl-L-carnitine Hydrochloride)) vs Arm II (Placebo); Test type: Superiority; p = 0.46, Regression, Linear; Adjusted for randomization stratification factors

5. Other Pre Specified Outcome: Serum Nerve Growth Factor Levels
Time Frame: 12 weeks post-registration
Population: Data still in process; Analysis to be performed in future.
Arm/Group | Arm I (Acetyl-L-carnitine Hydrochloride)) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Treatment and Concurrent Therapy
Description: total dose of taxane received and treatment delays, compliance with therapy, and use of concurrent medications, dietary supplements (e.g., glutamine), vitamin E, and complementary and alternative medicines
Time Frame: 12 weeks post-registration
Population: Data still in process; Analysis to be performed in future.
Arm/Group | Arm I (Acetyl-L-carnitine Hydrochloride)) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Association Between Nerve Growth Factor Levels and the Degree of Neuropathy and Functional Status
Description: Explore the relationship between nerve growth factor levels and the degree of neuropathy and functional status in these patients.
Time Frame: 12 weeks post-registration
Population: Data still in process; Analysis to be performed in future.
Arm/Group | Arm I (Acetyl-L-carnitine Hydrochloride)) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Association Between Genetic Markers Responsible for Taxane Metabolism and Clearance and the Degree of Neuropathy
Description: Explore the relationship between genetic markers responsible for taxane metabolism and clearance (e.g., CYP2C8, CYP3A4, CYP3A5, GSTM1, and GSTP1) and the degree of neuropathy in these patients.
Time Frame: 12 weeks post-registration
Population: Data still in process; Analysis to be performed in future.
Arm/Group | Arm I (Acetyl-L-carnitine Hydrochloride)) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 25 weeks
Arm/Group | Arm I (Acetyl-L-carnitine Hydrochloride)) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 1/208 | 0/201
Other Adverse Events (participants affected / at risk) | 156/208 | 153/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Acetyl-L-carnitine Hydrochloride)) (N=208) | Arm II (Placebo) (N=201)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Acetyl-L-carnitine Hydrochloride)) (N=208) | Arm II (Placebo) (N=201)
Diarrhea (Gastrointestinal disorders) | 13 | 10
Nausea (Gastrointestinal disorders) | 46 | 51
Vomiting (Gastrointestinal disorders) | 17 | 14
Fatigue (asthenia, lethargy, malaise) (General disorders) | 38 | 32
Pain - Joint (Musculoskeletal and connective tissue disorders) | 13 | 12
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 12 | 9
Neuropathy: motor (Nervous system disorders) | 18 | 16
Neuropathy: sensory (Nervous system disorders) | 127 | 127
Insomnia (Psychiatric disorders) | 51 | 45
Hot flashes/flushes (Vascular disorders) | 21 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No